CLINICAL TRIAL: NCT04226482
Title: Comparison of Lateral Thermal Damage and Clinical Outcomes of Laparoscopic Appendectomy With New Versus Reused Ultrasonic Scalpel in Patients With Acute Appendicitis - Randomized Clinical Trial
Brief Title: Review of Efficacy of Used ultraSonic Energy Device
Acronym: REUSED
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Split, School of Medicine (Other)
Collaborators: University Hospital of Split (Other); General Hospital Zadar (Other)
Responsible Party: Principal Investigator, Jakov Mihanovic, Jakov Mihanovic, Principal Investigator, University of Split, School of Medicine
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REUSED2019
Record Dates: First submitted 2019-12-28; First posted 2020-01-13 (Actual); Last update posted 2020-05-18 (Actual); Status verified 2020-05

CONDITIONS: Appendicitis Acute; Safety Issues; Complication of Surgical Procedure; Device Induced Injury
Keywords: Appendectomy; Laparoscopic Surgery; Equipment Reuse; Patient Safety
MeSH Terms: conditions — Appendicitis | interventions — Device Approval

STUDY DESIGN:
Intervention Model Description: Participants will be randomized to laparoscopic appendectomy with new ultrasonic shears versus laparoscopic appendectomy with reused ultrasonic shears. Randomization sequence will be issued by independent statistician and the participants will be blinded to the surgical instrument used for laparoscopic appendectomy.
Who Masked: Participant
Masking Description: Participants will be blinded to allocation and instrument used for surgery, with the same clinical treatment and postoperative follow-up.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- New Device (Active Comparator): Laparoscopic appendectomy will be done using new ultrasonic shears.
  Interventions: Device: New Device
- Used Device (Experimental): Laparoscopic appendectomy will be done using reprocessed ultrasonic shears.
  Interventions: Device: Used Device

INTERVENTIONS:
Device: New Device — Laparoscopic appendectomy using new ultrasonic shears.
  Arms: New Device
Device: Used Device — Laparoscopic appendectomy using reprocessed ultrasonic shears.
  Arms: Used Device

SUMMARY:
Single-use medical instruments are intended by the manufacturers for single-use only or for single-patient-use only. Nevertheless, single-use instruments are being reused more than once in many countries around the world. The reasons are mainly economic in developing countries and environmental in developed countries. Concerns are being raised regarding reused instruments sterility and efficacy. Since there is paucity of evidence on safety of multiple use of single-use instruments in surgery, we decided to conduct a clinical study comparing the same surgical procedure performed with new versus reused surgical instrument. We decided to study laparoscopic appendectomy which is a simple and the most common emergency surgery. Instrument under the scrutiny is ultrasonic scalpel which uses high-frequency ultrasound vibration for coagulating and cutting tissue. In the studied period of time, all eligible patients with acute appendicitis will be randomized in two groups, first having surgery with new device and the second having surgery with reused device. Removed appendix will be analyzed for lateral thermal damage and the patients will be followed-up for one month for potential differences in clinical outcomes like pain-killers consumption, length of stay and postoperative complications.

DETAILED DESCRIPTION:
Laparoscopic appendectomy provides enhanced recovery at increased costs due to a need for a specific sophisticated equipment. Currently many of the commonly used devices are labeled by manufacturers as single-use only. This trend has stronghold in concerns about patient safety, especially about prevention of cross-infections and other safety-related issues. On the other hand, surgery costs are increased exponentially. There is paucity of evidence on safety of reusing single-use devices (SUD) in surgery. Reuse of SUD which may include refurbishing or reprocessing and resterilization is a complex issue with moral, technical, economical and environmental repercussions. There are several papers discussing the ethical dilemmas involved. The reprocessed instruments are generally deemed equally safe as new one. However there are only few experimental and clinical studies on this topic. Most of them are influenced by sponsors or manufacturers and therefore biased. What's more their conclusions are sometimes highly controversial. Goal of this study is to provide solid evidence on safety of reuse of SUD and to discover differences in in-vitro and clinical outcomes. One of the most common SUD for laparoscopic surgery is ultrasonic scalpel which uses high-frequency jaw vibration which simultaneously coagulates and divides structures with minimal thermal damage to surrounding tissue. One of the best known ultrasonic shears intended for single-use is harmonic scalpel (Ultracision® Ethicon EndoSurgery, Johnson&Johnson Company). Ultrasonic shears are being refurbished and/or resterilized for repetitive use in limited number of cycles or until become dysfunctional or disintegrate. Routine depends on local regulations and variations in practice. To encourage or to ban aforementioned practice we need solid evidence based on properly conducted clinical trial. Therefore we have designed a single-blind randomised clinical trial depending on virginity of instrument used for tissue dissection. Since Ultracision device is the most commonly used ultrasonic sealing device we decided to study outcomes of surgery performed with the new (unused) instrument versus resterilized reused instrument.

All of the patients with clinical and radiological suspicion of having acute appendicitis will be blindly allocated in two arms according to the predefined random sequence provided by independent statistician. Eligible patients will sign an informed consent form. First arm will have laparoscopic appendectomy with new ultrasonic device. The patient will be blinded for the allocation, but the surgeon can not be blinded since packing of the new and reused instruments differ. Even if the scrub nurse would give surgeon instruments without packing, some minor damage might be seen on the plastic coating of the instrument jaws. The second arm will have laparoscopic appendectomy with reused ultrasonic device. All other treatment including surgical technique, postoperative management and follow-up will be unchanged or within the standard of care. Surgical technique is standardised three-trocar approach in general anesthesia. All other details of the surgery are variable depending on local findings, extent of inflammation, anatomy variations etc. Removed specimens will be analyzed routinely with addition of measurement of lateral thermal damage of mesoappendix and appendiceal base. Patients will be screened for antibiotic therapy length, analgesics consumption, early surgical complications according to Clavien-Dindo classification and length of stay. Additionally one month follow-up will be conducted to pick-up possible late complications or readmissions. Study will be conducted in two centers for a period of time until sufficient number of participants are recruited.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of acute appendicitis confirmed during surgery
* Laparoscopic appendectomy
* Operated with UltraCision harmonic scalpel.

Exclusion Criteria:

* Finding of innocent (white) appendix
* Pregnancy
* Significant co-morbidity (ASA III-IV)
* Open appendectomy
* Laparoscopic appendectomy using instruments other than Ultracision harmonic scalpel.

Ages: 5 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2019-05-27 (Actual); Primary Completion 2020-04-13 (Actual); Study Completion 2020-05-14 (Actual)

PRIMARY OUTCOMES:
Lateral Thermal Damage of Mesoappendix | Through study completion, an average of 1 year.
  Microscopically measured distance of lateral thermal damage of mesoappendix
Lateral Thermal Damage of Appendiceal Base | Through study completion, an average of 1 year.
  Microscopically measured distance of lateral thermal damage of appendiceal base

SECONDARY OUTCOMES:
Clinical outcome - Postoperative complications | Postoperative 30 days follow-up
  Clavien Dindo classification of postoperative complications
Clinical outcome - Length of stay | Through study completion, an average of 1 year.
  In-hospital stay in days
Time to transect appendiceal base | During the surgery
  Speed of transection of appendiceal base regarding its diameter in seconds
Rating Device Functionality | Immediately after surgery
  Rating of Surgeon's satisfaction with ultrasonic shears' performance using Performance Evaluation Scale (PES) where: 1 is unacceptable, 2 is acceptable, 3 is optimal.
  PES has 5 categories: 1. Hemostasis, 2. Coagulation effect, 3. Cutting effect, 4. Instrument activation force, 5. Disturbing sounds.

CONTACTS AND LOCATIONS:
Overall Officials: Jakov Mihanovic, MD, Principal Investigator — General Hospital Zadar
Locations (2):
- Croatia (2):
  - Clinical Hospital Split, Split
  - General Hospital Zadar, Zadar

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chu T, Chandhoke RA, Smith PC, Schwaitzberg SD. The impact of surgeon choice on the cost of performing laparoscopic appendectomy. Surg Endosc. 2011 Apr;25(4):1187-91. doi: 10.1007/s00464-010-1342-1. Epub 2010 Sep 11. PMID 20835717
- [Background] Dunn D. Reprocessing single-use devices--the ethical dilemma. AORN J. 2002 May;75(5):989-99; quiz 1000-4. doi: 10.1016/s0001-2092(06)61462-2. PMID 12063946
- [Background] Collier R. The ethics of reusing single-use devices. CMAJ. 2011 Aug 9;183(11):1245. doi: 10.1503/cmaj.109-3907. Epub 2011 Jul 11. No abstract available. PMID 21746819
- [Background] Lester BR, Miller K, Boers A, Harris DC, Gamble WG. Comparison of in vivo clinical performance and shaft temperature and in vitro tissue temperature and transection times between new and reprocessed harmonic scalpels. Surg Laparosc Endosc Percutan Tech. 2010 Oct;20(5):e150-9. doi: 10.1097/SLE.0b013e3181eff973. PMID 20975490
- [Background] Weld KJ, Dryer S, Hruby G, Ames CD, Venkatesh R, Matthews BD, Landman J. Comparison of mechanical and in vivo performance of new and reprocessed harmonic scalpels. Urology. 2006 May;67(5):898-903. doi: 10.1016/j.urology.2005.11.027. PMID 16698349
- [Background] Jacobs P, Akpinar I. Single-use medical devices: economic issues. Heart Asia. 2018 Nov 9;10(2):e011034. doi: 10.1136/heartasia-2018-011034. eCollection 2018. No abstract available. PMID 30556542
- [Background] Hailey D, Jacobs PD, Ries NM, Polisena J. Reuse of single use medical devices in Canada: clinical and economic outcomes, legal and ethical issues, and current hospital practice. Int J Technol Assess Health Care. 2008 Fall;24(4):430-6. doi: 10.1017/S0266462308080562. PMID 18828937
- [Background] Sloan TW. Safety-cost trade-offs in medical device reuse: a Markov decision process model. Health Care Manag Sci. 2007 Feb;10(1):81-93. doi: 10.1007/s10729-006-9007-2. PMID 17323656
- [Background] Collier R. Reprocessing single-use devices: an international perspective. CMAJ. 2011 Aug 9;183(11):1244. doi: 10.1503/cmaj.109-3906. Epub 2011 Jul 4. No abstract available. PMID 21727228
- [Background] Popp W, Rasslan O, Unahalekhaka A, Brenner P, Fischnaller E, Fathy M, Goldman C, Gillespie E. What is the use? An international look at reuse of single-use medical devices. Int J Hyg Environ Health. 2010 Jul;213(4):302-7. doi: 10.1016/j.ijheh.2010.04.003. Epub 2010 May 13. PMID 20471316
- [Background] Magetsari R, van der Houwen EB, Bakker MT, van der Mei HC, Verkerke GJ, Rakhorst G, Hilmy CR, van Horn JR, Busscher HJ. Biomechanical and surface physico-chemical analyses of used osteosynthesis plates and screws--potential for reuse in developing countries? J Biomed Mater Res B Appl Biomater. 2006 Nov;79(2):236-44. doi: 10.1002/jbm.b.30534. PMID 16680715
- [Background] Roth K, Heeg P, Reichl R. Specific hygiene issues relating to reprocessing and reuse of single-use devices for laparoscopic surgery. Surg Endosc. 2002 Jul;16(7):1091-7. doi: 10.1007/s00464-001-9190-7. Epub 2002 Apr 9. PMID 12165829
- [Background] Fengler TW, Pahlke H, Bisson S, Kraas E. The clinical suitability of laparoscopic instrumentation. A prospective clinical study of function and hygiene. Surg Endosc. 2000 Apr;14(4):388-94. doi: 10.1007/s004640020064. PMID 10790561
- [Background] Manatakis DK, Georgopoulos N. Reducing the Cost of Laparoscopy: Reusable versus Disposable Laparoscopic Instruments. Minim Invasive Surg. 2014;2014:408171. doi: 10.1155/2014/408171. Epub 2014 Jul 22. PMID 25152814
- [Background] Druzijanic N, Pogorelic Z, Perko Z, Mrklic I, Tomic S. Comparison of lateral thermal damage of the human peritoneum using monopolar diathermy, Harmonic scalpel and LigaSure. Can J Surg. 2012 Oct;55(5):317-21. doi: 10.1503/cjs.000711. PMID 22854112
- [Background] Pogorelic Z, Katic J, Mrklic I, Jeroncic A, Susnjar T, Jukic M, Vilovic K, Perko Z. Lateral thermal damage of mesoappendix and appendiceal base during laparoscopic appendectomy in children: comparison of the harmonic scalpel (Ultracision), bipolar coagulation (LigaSure), and thermal fusion technology (MiSeal). J Surg Res. 2017 May 15;212:101-107. doi: 10.1016/j.jss.2017.01.014. Epub 2017 Jan 28. PMID 28550895
- [Background] Zilberstein. Reprocessamento de pincas de alta resolucao para corte e coagulacao. ABCD Arq Bras Cir Dig. 2013.
- [Background] Colak T, Ersoz G, Akca T, Kanik A, Aydin S. Efficacy and safety of reuse of disposable laparoscopic instruments in laparoscopic cholecystectomy: a prospective randomized study. Surg Endosc. 2004 May;18(5):727-31. doi: 10.1007/s00464-004-8112-x. Epub 2004 Mar 19. PMID 15026911
- [Background] Ramshaw BJ. Reusing disposal laparoscopic instruments. Surg Endosc. 2004 Aug;18(8):1161-2. doi: 10.1007/s00464-004-8203-8. Epub 2004 Jul 7. No abstract available. PMID 15457375
- [Background] Chan AC, Ip M, Koehler A, Crisp B, Tam JS, Chung SC. Is it safe to reuse disposable laparoscopic trocars? An in vitro testing. Surg Endosc. 2000 Nov;14(11):1042-4. doi: 10.1007/s004640000118. PMID 11116415
- [Background] DesCoteaux JG, Tye L, Poulin EC. Reuse of disposable laparoscopic instruments: cost analysis. Can J Surg. 1996 Apr;39(2):133-9. PMID 8769924
- [Background] Emam TA, Cuschieri A. How safe is high-power ultrasonic dissection? Ann Surg. 2003 Feb;237(2):186-91. doi: 10.1097/01.SLA.0000048454.11276.62. PMID 12560776
- [Background] Lopes Cde L, Graziano KU, Pinto Tde J. Evaluation of single-use reprocessed laparoscopic instrument sterilization. Rev Lat Am Enfermagem. 2011 Mar-Apr;19(2):370-7. doi: 10.1590/s0104-11692011000200020. English, Portuguese, Spanish. PMID 21584385
- [Background] Mues AC, Haramis G, Casazza C, Okhunov Z, Badani KK, Landman J. Prospective randomized single-blinded in vitro and ex vivo evaluation of new and reprocessed laparoscopic trocars. J Am Coll Surg. 2010 Dec;211(6):738-43. doi: 10.1016/j.jamcollsurg.2010.08.003. Epub 2010 Oct 30. PMID 21036630
- [Background] Gartner D, Munz K, Huckelheim E, Hesse U. [Ultrasonic scissors. New vs resterilized instruments]. Chirurg. 2008 Feb;79(2):175-9. doi: 10.1007/s00104-007-1420-7. German. PMID 18259794
- [Background] Bruning LM. Disposables v. reusables in OR practice: Part I, Weighing contributions to patient care. Nurs Manage. 1992 Feb;23(2):80J-80K, 80N, 80P. doi: 10.1097/00006247-199202000-00026. No abstract available. PMID 1736216
- [Background] Bruning LM. Disposables v. reusables in or practice: Part II, Weighing costs, risks and wastes. Nurs Manage. 1992 Mar;23(3):72I-72K, 72N, 72P. doi: 10.1097/00006247-199203000-00024. No abstract available. PMID 1553152
- [Background] Uyeno et al. Experimental study on the analysis of sterility in the reuse of harmonic scalpels. Revista Brasileira de Ciencias Medicas e da Saude (Brazilian J Medical Science and Health). 2015.
- [Background] Kadesky KM, Schopf B, Magee JF, Blair GK. Proximity injury by the ultrasonically activated scalpel during dissection. J Pediatr Surg. 1997 Jun;32(6):878-9. doi: 10.1016/s0022-3468(97)90641-2. PMID 9200091
- [Background] Kinoshita T, Kanehira E, Omura K, Kawakami K, Watanabe Y. Experimental study on heat production by a 23.5-kHz ultrasonically activated device for endoscopic surgery. Surg Endosc. 1999 Jun;13(6):621-5. doi: 10.1007/s004649901055. PMID 10347305
- [Background] Klar M, Haberstroh J, Timme S, Fritzsch G, Gitsch G, Denschlag D. Comparison of a reusable with a disposable vessel-sealing device in a sheep model: efficacy and costs. Fertil Steril. 2011 Feb;95(2):795-8. doi: 10.1016/j.fertnstert.2010.09.014. Epub 2010 Oct 16. PMID 20951375
- [Background] Laustsen G. Reduce--recycle--reuse: guidelines for promoting perioperative waste management. AORN J. 2007 Apr;85(4):717-22, 724, 726-8. doi: 10.1016/S0001-2092(07)60146-X. PMID 17418129
- [Background] Gartner D, Munz K, Huckelheim E, Hesse U. Ultrasound scissors: new single-use instruments vs. resterilised single-use instruments - a prospective randomised study. GMS Krankenhhyg Interdiszip. 2008 Sep 3;3(3):Doc20. PMID 20204092
- [Background] Yung E, Gagner M, Pomp A, Dakin G, Milone L, Strain G. Cost comparison of reusable and single-use ultrasonic shears for laparoscopic bariatric surgery. Obes Surg. 2010 Apr;20(4):512-8. doi: 10.1007/s11695-008-9723-4. Epub 2008 Nov 18. PMID 19015932
- [Background] Siu J, Hill AG, MacCormick AD. Systematic review of reusable versus disposable laparoscopic instruments: costs and safety. ANZ J Surg. 2017 Jan;87(1-2):28-33. doi: 10.1111/ans.13856. Epub 2016 Nov 23. PMID 27878921
- [Background] Hussain M, Balsara KP, Nagral S. Reuse of single-use devices: looking back, looking forward. Natl Med J India. 2012 May-Jun;25(3):151-5. PMID 22963293
- [Background] Renton D, Denk P, Varban O. Reprocessed single-use devices in laparoscopy: assessment of cost, environmental impact, and patient safety. Surg Endosc. 2018 Oct;32(10):4310-4313. doi: 10.1007/s00464-018-6275-0. Epub 2018 Jun 15. No abstract available. PMID 29905894
- [Background] Jacobs P, Polisena J, Hailey D, Lafferty S. Economic analysis of reprocessing single-use medical devices: a systematic literature review. Infect Control Hosp Epidemiol. 2008 Apr;29(4):297-301. doi: 10.1086/529587. PMID 18462140
- [Background] Martins et al. Reprocessing of single-use medical devices: clinical and financial results. Port J Public Health. 2019.
- [Background] Brady JT, Bhakta A, Steele SR, Trunzo JA, Senagore AJ, Holmgren K, Schillero A, Champagne BJ. Reprocessed bipolar energy for laparoscopic colectomy: Is it worth it? Am J Surg. 2017 Jul;214(1):59-62. doi: 10.1016/j.amjsurg.2017.02.012. Epub 2017 Feb 20. PMID 28279396
- [Derived] Mihanovic J, Sikic NL, Mrklic I, Katusic Z, Karlo R, Jukic M, Jeroncic A, Pogorelic Z. Comparison of new versus reused Harmonic scalpel performance in laparoscopic appendectomy in patients with acute appendicitis-a randomized clinical trial. Langenbecks Arch Surg. 2021 Feb;406(1):153-162. doi: 10.1007/s00423-020-02039-y. Epub 2020 Nov 25. PMID 33241426
- See also: The Reprocessing and Reuse of Single-Use Medical Devices in Newfoundland & Labrador (2010) — https://www.nlcahr.mun.ca/CHRSP/SUDS_full_web.pdf
- See also: Safety and performance evaluation of remanufactured harmonic scalpels (2010) — http://www.amdr.org/wp-content/uploads/2010/09/White-Paper-Safety-and-Performance-Eval-of-Remfd-Harmonic-Scalpels.pdf
- See also: Croatian Law on Medical Products 2017/745 (2018) - Article in Croatian — https://www.zakon.hr/z/1253/Zakon-o-provedbi-Uredbe-%28EU%29-2017-745-o-medicinskim-proizvodima-i-Uredbe-%28EU%29-2017-746-o-in-vitro-dijagnostičkim-medicinskim-proizvodima